CLINICAL TRIAL: NCT02215187
Title: Cognitive Behavioral Therapy (CBT) for Caregivers of Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) Service Members With Combat-Related Traumatic Brain Injuries (TBI)
Brief Title: Telehealth-Education-Based Program for Military Caregivers of Injured Service Members With Head Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura E. Dreer, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #000435754; H133G110275 (Other Grant/Funding Number: NIDRR/H133G110275)
Record Dates: First submitted 2014-06-24; First posted 2014-08-13 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem-Solving Training (Experimental): PST is a cognitive-behavioral intervention. Delivery of the PST + usual care condition will be administered to caregivers over the course of 6 one-hour per week, telephone calls/sessions that will entail education related to problem-solving skills/problem-solving model and application to caregiving and managing caregiver related problems.
  Interventions: Behavioral: Problem-Solving Training (PST)
- Attention Control (Sham Comparator): Attention/social contact control. Health education (non-skill focused).
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Problem-Solving Training (PST) — Training in problem-solving skills to be applied to military caregiver problems.
  Arms: Problem-Solving Training
Behavioral: Attention Control — Social contact control (health education/no skill training)
  Other Names: Social contact control
  Arms: Attention Control

SUMMARY:
The primary purpose of this research is to evaluate the impact of a telehealth-based, cognitive behavioral therapy (CBT) intervention (problem-solving training: PST) for adult informal military family/friend caregivers of OIF/OEF service members with a deployment-related TBI.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) has gained increasing attention in American society as it is now considered the "signature injury" of the Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF) campaigns. The chronic changes that often occur in the wake of TBI along with possible physical injuries may run a chronic, unremitting course, imposing great strain and distress upon family members who often assume a caregiver role with little preparation and no formal training for these wounded service members as they reintegrate back into civilian life post-deployment. Unfortunately, research has not adequately addressed the unique long-term needs of informal military caregivers of deployed service members with TBI (i.e., family members/close friends).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years old
* Meets study project definition of a military caregiver
* Documentation or determination of an OIF/OEF deployment related TBI
* Service member will have presented to a Veterans Administration Medical Center (VAMC) or military medical center
* English-speaking
* Has access to a telephone for the administration of measures and/or intervention calls
* Has no significant cognitive or communication problems that might significantly interfere with adequately understanding information or talking on the telephone which will be determined by the clinical judgment of the person consenting the participant.

Exclusion Criteria:

* Has a life-threatening or other serious disease that impacts the ability to participate for the duration of the project
* No determination or documentation of a deployment-related TBI related to OIF/OEF for the injured service member
* Has a severe hearing impairment that impedes communication and standardized implementation of the intervention and telephone follow-up
* Formal caregiver
* Caregiver does not want to participate

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | Change from baseline in PHQ-9 scores at post-program (3-months follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dreer, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States